CLINICAL TRIAL: NCT03903315
Title: Central Malignant Airway Obstructions: Medical Treatment Alone Versus Endoscopic and Medical Treatment. A Multicentric Retrospective Study
Brief Title: Central Malignant Airway Obstructions: Medical Treatment Alone Versus Endoscopic and Medical Treatmen
Acronym: EVERMORE
Status: Completed | Type: Observational
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Alessandro Marchioni, Principal Investigator, University of Modena and Reggio Emilia
Other Study IDs: UModenaReggio 7
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Endobronchial Mass; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- medical treatment alone: Patients with central malignant airway obstructions undergoing medical treatment alone
  Interventions: Other: Comparison between patients with Patients with central malignant airway obstructions undergoing medical treatment alone versus medical and endoscopic treatment
- endoscopic + medical treatment: Patients with central malignant airway obstructions undergoing medical and endoscopic treatment
  Interventions: Other: Comparison between patients with Patients with central malignant airway obstructions undergoing medical treatment alone versus medical and endoscopic treatment

INTERVENTIONS:
Other: Comparison between patients with Patients with central malignant airway obstructions undergoing medical treatment alone versus medical and endoscopic treatment — Comparison between patients with Patients with central malignant airway obstructions undergoing medical treatment alone versus medical and endoscopic treatment with reference to mortality and complications.

SUMMARY:
The obstruction of the central airways (CAO) may be caused by a large variety of malignant and non malignant processes, and it may present with a variety of symptoms ranging from mild shortness of breath to life-threatening respiratory failure.

The epidemiologic impact of lung cancer leads to an increasing number of patients developing complications of proximal endobronchial disease. An estimated 20-30% of patients with lung cancer will develop complications associated with airway obstruction, e.g. dyspnea, pneumonia and atelectasis, and up to 40% of lung cancer deaths may be attributed to locoregional disease.

Although lung cancer patients with CAO are not candidates for surgical resection, more than 80% of these patients can receive palliative treatment using interventional bronchoscopy; in addiction, almost the 85% of these procedures reach luminal clearance and endoscopic success in terms of symptomatic relief, of pulmonary function and quality of life.

There are no definitive data about factors such as type of disease or site of the lesion which may affect the use of a single or a combined endoscopic modality or stenting in the treatment of airway obstructions. A Dalar's retrospective study showed that airway stenting is a useful treatment modality besides the other interventional bronchoscopic procedures: it not only provides rapid relief of symptoms and an improved quality of life, but also gives additional time for adjuvant chemo-radiotherapy that might provide prolonged survival.

Since Dumon introduced the first dedicated endoluminal airway stent, there was a clear immediate relief of respiratory symptoms and significant quality survival in most patients (9). In a Miyazawa's study all patients with malignant central airway obstruction had significant improvements in dyspnea and also in spirometry after stenting, and the author suggested that the correct positioning of the stent at the choke point leads to maximal symptomatic benefit in these patients. The choice of different airway stents can be made based on the nature (intrinsic, extrinsic or combined) and site of the lesion: for example the Dumon stent can be preferred in lesions of trachea and right main bronchus, the Ultraflex stent on the left and stenosis beyond the main bronchi. The underlying disease, the site of lesion and treatment modality are known as independent predictors of survival. Complications related to the placement of stents include re-obstructions of the lumen by tumor, granuloma formation at the stent side, mucous plugging and migration of the stent; with the use of laser, both perforation of airway wall and fire.

Regarding laser resection for malignant airway obstruction, it is associated with improved survival rates (60% of patients alive at 7 months in one study). As these studies were not randomized trials, it is impossible to conclude that the laser therapy was responsible for the improved survival, but it is likely that laser therapy provided a rapid and safe means of relieving central airway obstruction, which is associated with a high mortality rate.

The strategy and modality of treatment for malignant central airway obstructions depends not only on the endoscopic characteristics and location of the lesions, but also on the patient's comorbidities, pulmonary function, previous treatment and life expectancy. The primary purpose of treatment with interventional bronchoscopy alone remains to improve symptom control and quality of life, not to improve the prognosis. However, the advent of molecular-targeted therapy may change the impact of interventional bronchoscopy, especially in lung cancer patients with EGFR mutations: in a Tomoyuki case report there is the first description of the use of endoscopic treatment plus molecular-targeted therapy as combination treatment, with benefits in terms of patient's general conditions and quality of life. Moreover, some researchers have reported cases of malignant lymphoma patients with central airway obstruction who were successfully treated using interventional bronchoscopy followed by systemic chemotherapy.

The aim of this study is to evaluate the differences between patients with central malignant airway obstruction treated only with medical therapy versus patients submitted to endoscopic plus medical therapy in terms of prognosis, quality of life and access to health services.

ELIGIBILITY:
Inclusion Criteria:

* patients with malignant central airways obstruction admitted to the Bronchoscopy Unit of the University Hospital of Modena (Italy) and to the Bronchoscopy Unit of the Arcispedale Santa Maria Nuova of Reggio Emilia (Italy)

Exclusion Criteria:

* metastatic disease
* small cell lung cancer
* pregnancy
* low performance status at the time of diagnosis

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with malignant central airways obstruction treated with medical therapy alone or endoscopic treatment and medical therapy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
1 year Survival | Ten years
  Assessment of survival through medical records and reports consultation

SECONDARY OUTCOMES:
Infections | Ten years
  Assessment of the onset of infections through medical records and reports consultation
Respiratory failure | Ten years
  Assessment of the onset of respiratory failure through medical records and reports consultation
Hospital admission | Ten years
  Assessment of the occurrence of hospital admission through medical records and reports consultation
Need for palliative care | Ten years
  Assessment of the need to start palliative support through medical records and reports consultation
Atelectasis | Ten years
  Assessment of the occurrence of atelectasis through medical records and reports consultation

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Policlinico di Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: Undecided